CLINICAL TRIAL: NCT03236220
Title: Effect of the Prophylactic Intervention of N-acetyl-L-cysteine (NAC) on the Incidence of Poor Graft Function and Prolonged Isolated Thrombocytopenia in Acute Leukemia Patients After Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Effect of NAC on the Hematopoietic Reconstitution After Haploidentical Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015PHB220
Record Dates: First submitted 2017-07-23; First posted 2017-08-01 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Haploidentical Hematopoietic Stem Cell Transplantation
Keywords: haploidentical hematopoietic stem cell transplantation; poor graft function; prolonged isolated thrombocytopenia; bone marrow endothelial cells; N-acetyl-L-cysteine; Acute leukemia
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-acetyl-L-cysteine group (Experimental): Acute leukemia patients with complete remission, whose bone marrow endothelial cells were less than 0.1% detected before haploidentical hematopoietic stem cell transplantation, receive N-acetyl-L-cysteine.
  Interventions: Drug: N-acetyl-L-cysteine

INTERVENTIONS:
Drug: N-acetyl-L-cysteine — Acute leukemia patients with complete remission, whose bone marrow endothelial cells were less than 0.1% detected before haploidentical hematopoietic stem cell transplantation, receive N-acetyl-L-cysteine (NAC) (orally at dosages of 400mg 3 times per day). NAC treatment begins from 14 days pre-allotransplant to 2 months after-allotransplant continuously in the absence of disease progression or unacceptable toxicity.
  Other Names: NAC

SUMMARY:
The aim of the study is to evaluate the efficacy of the prophylactic administration of N-acetyl-L-cysteine (NAC) in acute leukemia patients with complete remission pre- and post-allotransplant on the occurrence of poor graft function (PGF) and prolonged isolated thrombocytopenia (PT) after haploidentical hematopoietic stem cell transplantation. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective treatment of malignant hematopoietic diseases. However, the delayed hematopoietic reconstitution, including PGF and PT, remain serious complication after allo-HSCT, and the effective therapeutic strategies are limited. In murine studies, endothelial cells have been identified as a key cellular component supporting hematopoietic stem cells in the bone marrow microenvironment. Our previous prospective nested case-control study suggested that the frequency of bone marrow endothelial cells was markedly reduced in patients with PGF or PT. Moreover, our recent study further identified reduced bone marrow endothelial cells (<0.1%) pre-allotransplant was associated with significant higher incidences of PGF or PT after allo-HSCT. In addition, NAC treatment in vitro could quantitatively and functionally improve bone marrow endothelial cells derived from the patients with PGF or PT. Therefore, bone marrow endothelial cells (<0.1%) pre-allotransplant can be used to identify patients with a higher incidence of PGF or PT to provide timely prophylactic intervention of NAC to prevent the occurrence of delayed hematopoietic reconstitution post-transplant. The study hypothesis: Prophylactic intervention of NAC pre- and post-allotransplant could reduce the incidence of PGF and PT in acute leukemia patients after haploidentical hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Acute leukemia patients with complete remission, whose bone marrow endothelial cells were less than 0.1% detected before haploidentical hematopoietic stem cell transplantation, receive NAC (orally at dosages of 400mg 3 times per day). NAC treatment begins from 14 days pre-allotransplant to 2 months after-allotransplant continuously in the absence of disease progression or unacceptable toxicity. The effect of NAC on hematopoietic stem cells, megakaryocytes, immunologic subsets, and the elements of bone marrow microenvironment will be monitored pre- and post-allotransplant.

Drug：N-acetyl-L-cysteine (NAC) is orally administrated at dosages of 400mg 3 times per day. NAC treatment begins from 14 days pre-allotransplant to 2 months after-allotransplant continuously in the absence of disease progression or unacceptable toxicity.

Participant：Acute leukemia patients with CR, whose bone marrow endothelial cells were less than 0.1% detected before haploidentical hematopoietic stem cell transplantation.

Eligibility Ages Eligible for Study: 15-60 Years Genders Eligible for Study: Both Accepts The trial will be terminated in following situation

1. Severe toxicity occurrence
2. Cumulative incidence of relapse increased) (≥ 30%)
3. Cumulative incidence of mortality increased (≥ 30%)
4. Cumulative incidence of severe graft-versus-host disease increased (≥ 30%)

ELIGIBILITY:
Inclusion Criteria:

Acute leukemia patients with complete remission, whose bone marrow endothelial cells were less than 0.1% detected before haploidentical hematopoietic stem cell transplantation；

Exclusion Criteria:

1. Bronchial asthma;
2. Allergic to N-acetyl-L-cystein

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of poor graft function and prolonged isolated thrombocytopenia | Participants will be followed for 2 months post-HSCT.
  Number of participants with poor graft function and prolonged isolated thrombocytopenia will be calculated at 2-month post-HSCT.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events will be assessed by CTCAE v4.0 during oral administration of NAC. | From 14 days pre-HSCT to 2 months post-HSCT.
  Participants will be closely observed for NAC-related toxicities during the NAC administration until 2-month post-HSCT.
Effect of NAC on hematopoietic stem cells, megakaryocytes and the elements of bone marrow microenvironment. | Participants will be followed for 100 days post-HSCT.
  Examine hematopoietic stem cells, megakaryocytes and the elements of bone
  marrow microenvironment by flow cytometry and bone marrow histological examination.
Incidence of GVHD | Participants will be followed for 100 days post-HSCT.
  Number of participants with I-IV aGVHD will be observed for 100 days post-HSCT.
Incidence of relapse | Participants will be followed for 1 year post-HSCT.
  Number of participants with morphologic relapse will be calculated at one year post-HSCT.
Incidence of viral infection | Participants will be followed for 100 days post-HSCT.
  Number of participants with viral infection(CMV,EBV,et al) will be observed for 100 days post-HSCT.
Non-relapse mortality | Participants will be followed for 1 year post-HSCT.
  Number of participants with non-relapse mortality will be observed for 1 year post-HSCT.
Progression-free survival | Participants will be followed for 1 year post-HSCT.
  Number of participants survived with progression-free will be observed for 1 year post-HSCT.
Overall survival | Participants will be followed for 1 year post-HSCT.
  Number of participants survived for 1 year post-HSCT will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijng, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kong Y, Wang Y, Zhang YY, Shi MM, Mo XD, Sun YQ, Chang YJ, Xu LP, Zhang XH, Liu KY, Huang XJ. Prophylactic oral NAC reduced poor hematopoietic reconstitution by improving endothelial cells after haploidentical transplantation. Blood Adv. 2019 Apr 23;3(8):1303-1317. doi: 10.1182/bloodadvances.2018029454. PMID 31015207